CLINICAL TRIAL: NCT06722638
Title: Virtual Reality During Lumbar Punctures in Acute Lymphoblastic Leukemia
Acronym: VIRALL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Rally Foundation for Childhood Cancer Research (Other)
Responsible Party: Principal Investigator, Jennifer Levine, Medical Director, Survivorship and Supportive Care, Children's National Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000820
Record Dates: First submitted 2024-07-02; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
Keywords: Virtual Reality; Lumbar Puncture
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR Arm (Experimental): Pain and anxiety management in this arm will include: topical numbing cream 30 minutes prior to the scheduled procedure, option for a 0.05mg/kg (max 2 mg) oral/IV dose of lorazepam. VR headsets will be donned. After sterile cleaning of the lumbar spine area, lidocaine will be injected between L3-4 or L4-5 for local anesthetic. A 22-gauge needle of appropriate length (1.5, 2.5, 3.5 inch) will be used to access the intrathecal space. Cerebral spinal fluid will be collected for evaluation (standard procedure) and IT chemotherapy will be administered.
  Interventions: Other: Use of Virtual Reality Headset
- GA Arm (No Intervention): Pain and anxiety in this arm will be managed with general anesthesia, usually propofol, which is the current standard of care at Children's National Hospital.

INTERVENTIONS:
Other: Use of Virtual Reality Headset — Virtual Reality Headsets will be used to augment pain and anxiety management during therapeutic LPs in children with acute lymphoblastic leukemia
  Arms: VR Arm

SUMMARY:
Over 90% of children and adolescents diagnosed with acute lymphoblastic leukemia (ALL) will survive long term. Part of the successful treatment that patients receive is the delivery of chemotherapy directly into their spinal fluid via a spinal tap. This takes place approximately 20 times over the course of treatment. Most children and adolescents receive general anesthesia during this procedure to manage pain and anxiety. It is now understood that general anesthesia contributes to impairments in brain functioning in the long term. Therefore, it is important to identify ways to manage pain and anxiety during these procedures that does not include general anesthesia. The investigators propose to test whether virtual reality (VR: a technology that provides immersive experiences utilizing content uploaded on a headset), used with local anesthesia and the option for an anti-anxiety medication will be an adequate replacement for general anesthesia for participants 7 years of age and over, with ALL in the maintenance phase of treatment.

DETAILED DESCRIPTION:
Over 90% of children and adolescents diagnosed with acute lymphoblastic leukemia (ALL) will be long-term survivors. To help prevent disease recurrence in the central nervous system, patients receive intrathecal chemotherapy, delivered via lumbar puncture, at least 20 times over the course of treatment. Although critical for cure, this component of treatment is a risk factor for neurocognitive impairments that can subsequently affect the daily living skills and academic achievement of survivors. It is now understood that the general anesthesia used to manage pain and anxiety during lumbar punctures also contributes to impairments in neurocognitive functioning. Recent studies have demonstrated that the use of general anesthesia can be decreased by using local anesthesia and offering oral or IV anxiolytic medications. The investigators propose that adding virtual reality (VR: a technology that provides immersive experiences utilizing content uploaded on a headset), to local anesthesia and the option for anxiolytics will be superior to using those medications alone. The investigators' aim in this study is to demonstrate the feasibility of using VR, in conjunction with local anesthesia and oral/IV anti-anxiety medications, in participants 7 years of age and older with ALL in the maintenance phase of treatment. The multi-disciplinary investigator team, which includes experts in pediatric oncology, survivorship, patient reported outcomes, VR technology and VR content, is uniquely suited to successfully develop, implement, and evaluate this strategy. The investigators' long-term objective is to create a scalable and sustainable alternative to general anesthesia that will adequately manage pain and anxiety without compromising neurocognitive function. By systematically working towards this long-term objective, the investigators seek to help survivors of childhood cancer lead happy, normal lives, free from acquired neurocognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosis of ALL or Lymphoma (as they receive the same therapy)
* In maintenance phase of treatment
* Still have 2 maintenance cycles planned
* Aged 7 and over
* Patient able to speak English
* Caregiver able to complete consent and study questionnaires in English or Spanish

Exclusion Criteria:

* Relapsed or refractory disease
* Previously required ultrasound guided LP procedure
* Already does LPs without anesthesia

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Feasibility | At time of Procedure
  Number of participants able to receive intrathecal chemotherapy while using Virtual Reality to augment local anesthesia and the option of an anxiolytic for management of pain and anxiety during the lumbar puncture procedure.

SECONDARY OUTCOMES:
Secondary Outcome: Acceptability | 1-3 months after first Lumbar Puncture
  Number of participants who, having successfully received intrathecal chemotherapy using Virtual Reality with local anesthesia and the option of an anxiolytic, choose to undergo the next procedrue under the same circumstances.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers will be able to request access.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting information will be available following publication and for the next 5 years.